CLINICAL TRIAL: NCT03972540
Title: Effect of a Mindful Eating Intervention on Weight Management in Overweight and Obese Postmenopausal Breast Cancer Survivors
Brief Title: Effect of Mindful Eating on Weight Management in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Elisabeth Lilian Pia Sattler, Ph.D., B.S. Pharm, Assistant Professor, University of Georgia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002818
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasm Female
Keywords: Obesity; Mindful eating; Postmenopausal breast cancer survivors; Weight management; Cardiovascular health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful eating intervention (Experimental): The mindful eating intervention was taught by a mindfulness-based stress reduction instructor certified by the Center of Mindfulness at the University of Massachusetts Medical School.
  Interventions: Behavioral: Mindful eating intervention

INTERVENTIONS:
Behavioral: Mindful eating intervention — A Mindful Eating Workshop™ workbook was used for standardization and reproducibility of these sessions. The group sessions were focused on teaching applied strategies to consume food with intention and attention and aimed at improving emotional relationships with food. Intervention sessions were held once a week in the evening for 2 hours per session over 8 weeks. The intervention was delivered in a large conference room on the University of Georgia campus. Participants were required to attend seven out of eight sessions. If participants missed a session, they met with the instructor 30 minutes before the beginning of the following week's session to receive individual instruction on content of the missed session.

SUMMARY:
This pilot study examined changes in anthropometric measures as a result of and feasibility/ acceptability of a mindful eating intervention for overweight and obese postmenopausal breast cancer survivors.

DETAILED DESCRIPTION:
Being overweight is associated with increased risk for chronic disease and premature death in breast cancer survivors. This pilot study examined changes in anthropometric measures as a result of and feasibility/ acceptability of a mindful eating intervention for overweight and obese postmenopausal breast cancer survivors. The one-group pre-posttest study design included eight weekly group-based mindful eating sessions on strategies to intentionally and attentively consume food. Anthropometrics, blood pressure, mindfulness, nutritional intake, and physical activity were collected at baseline and 12-weeks follow-up. Data on feasibility and acceptability were collected at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female
* Breast cancer survivor (in remission)
* Completed cancer treatment at the time of study enrollment
* Body Mass Index (BMI) equal or greater than 25 kg/m²

Exclusion Criteria:

* None.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Change measured between weeks 1 and 12
  At the baseline and follow-up visits, trained study staff measured participants' weight and height using a standardized protocol. Height (measured by a stadiometer to the nearest 0.1 cm) and weight (measured by a scale to the nearest 0.1 kg) was used to calculate BMI (weight in kg divided by height in m²).
Blood Pressure | Change measured between weeks 1 and 12
  At the baseline and follow-up visits, trained study staff measured participants' systolic/diastolic blood pressure using a standardized protocol to the nearest mmHg. In order to ensure reliability, all measurements were taken 3 times and average values were used for analyses.
Waste and Hip Circumference | Change measured between weeks 1 and 12
  At the baseline and follow-up visits, trained study staff measured participants' waist and hip circumference by tape measure to the nearest 0.1 centimeter.
Body Fat Percentage | Change measured between weeks 1 and 12
  At the baseline and follow-up visits, trained study staff measured participants' body fat percentage using a bioelectrical impedance analyzer (BIA).
Feasibility of Conducting the Intervention | Measured at week 12
  Feasibility was assessed by tracking participant accrual and retention rates.
Acceptability of the Intervention | Measured at week 12
  To measure acceptability, participants were asked to complete a 5-question feedback survey to evaluate the mindful eating intervention at the follow-up study visit. Specifically, the open-ended survey questions asked participants about (1) their experience with intervention, (2) how the intervention affected diet and exercise management, (3) positive aspects about the intervention, (4) negative aspects about the intervention, and (5) suggested changes to the intervention. Qualitative data analysis techniques were used to identify themes within the data.

SECONDARY OUTCOMES:
Mindful Eating Measures | Change measured between weeks 1 and 12
  Changes in mindfulness resulting from the intervention were measured using the validated Mindful Attention Awareness Scale (MAAS). The MAAS questionnaire is a 15-item scale that was designed to assess mindfulness and receptive awareness throughout an individual's daily life. Scores from the MAAS range from 1 to 6, with higher scores associated with higher mindfulness. The MAAS was validated for use in cancer populations against the Profile of Mood States (POMS) scale that is widely used in clinical settings. Higher MAAS scores were significantly correlated with lower POMS scores, further confirming the construct validity of the MAAS questionnaire for assessing mindfulness in cancer populations. The questionnaire was self-administered to the participants pre and post intervention.

OTHER OUTCOMES:
Nutritional Intake | Change measured between weeks 1 and 12
  Habitual nutritional intake was measured using an electronic version of the Block Food Frequency Questionnaire, a 127-item food and beverage recall instrument referencing the consumption over the past month. Dietary intake data was describes as daily energy consumption (kcal), consumption of macronutrients (fat, protein, carbohydrate; grams/day), and intake of sweets (% of daily intake) to compare intake before intervention start with intake during the intervention.
Physical Activity | Change measured between weeks 1 and 12
  Participants' physical activity levels (average daily steps; moderate-to-vigorous physical activity (MVPA) minutes) were tracked throughout the study period using FitBit® Flex accelerometers. Total daily steps and MVPA minutes were averaged for the first and the last week of the intervention to examine changes.

IPD SHARING:
Plan to Share IPD: No